CLINICAL TRIAL: NCT07310732
Title: Clinical and Tomographic Efficacy of the Modified Minimally Invasive Surgical Technique (M-MIST) Alone and Combined With Enamel Matrix Derivative (EMD) and Bone Mineral Derived Xenograft (BMDX), in the Treatment of Isolated, Inter-dental Intra-bony Defects
Brief Title: Clinical and Radiographic Assessment of Efficacy of Modified Minimally Invasive SurgicalTechnique (M-MIST) Alone and Combined With Enamel Matrix Proteins and Ox-derived Bone Graft in the Treatment of Single Bone Defects Between Teeth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rungta College of Dental Sciences and Research (Other)
Responsible Party: Principal Investigator, Karthik Krishna M, Dean, Rungta College of Dental Sciences and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCDSR/IEC/MDS/2021/b-11
Record Dates: First submitted 2025-09-26; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Diseases; Periodontal Bone Loss
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss | interventions — enamel matrix proteins; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- modified minimally invasive surgical technique (Placebo Comparator)
  Interventions: Procedure: modified minimally invasive surgical technique
- modified minimally invasive surgical technique with emdogain (Active Comparator)
  Interventions: Procedure: modified minimally invasive surgical technique plus emdogain
- modified minimally invasive surgical technique with emdogain and xenograft (Experimental)
  Interventions: Procedure: modified minimally invasive surgical technique plus emdogain and xenograft

INTERVENTIONS:
Procedure: modified minimally invasive surgical technique — modified minimally invasive surgical technique alone in interdental area
  Arms: modified minimally invasive surgical technique
Procedure: modified minimally invasive surgical technique plus emdogain — modified minimally invasive surgical technique with application of enamel matrix proteins in interdental area
  Arms: modified minimally invasive surgical technique with emdogain
Procedure: modified minimally invasive surgical technique plus emdogain and xenograft — modified minimally invasive surgical technique with application of enamel matrix proteins and placement of bovine bone graft in interdental area
  Arms: modified minimally invasive surgical technique with emdogain and xenograft

SUMMARY:
This study was performed to investigate the adjunctive clinical benefit of the application of enamel matric derivatives and xenograft with the modified minimally invasive surgical technique in the treatment of isolated intrabony defects in periodontally compromised subjects.

ELIGIBILITY:
Inclusion Criteria:

* at least one site associated with an intrabony defect of ≥3 mm involving predominantly the interdental space of the tooth
* patients with optimal compliance

Exclusion Criteria:

* Patients with uncontrolled or poorly controlled diabetes
* history of long-term use of medications
* allergic to medications
* pregnant or lactating women
* smokers/users of other tobacco products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | 24 weeks
  The depth of probe penetration into the pocket (millimeters) is measured from the gingival margin using an UNC-15 probe.
Clinical Attachment Level | 24 weeks
  The distance from the base of the pocket to cemento-enamel junction (millimeters) is measured using an UNC-15 probe.

SECONDARY OUTCOMES:
Full mouth plaque score | 24 weeks
  Turesky Modification of Quigley-Hein Index used to assess plaque buildup across all tooth surfaces (buccal, lingual, mesial, distal) with scoring 0 (no plaque) to 5 (heavy plaque)
Full mouth bleeding score | 24 weeks
  Probe is inserted and withdrawn at the distal point of the tooth and monitored for bleeding within 10 seconds. Registered with (+) availability of provoked bleeding and with (-) its absence.
Mean defect depth | 24 weeks
  measured as the distance fromt the alveolar crest to the base of the defect (in CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontics, Rungta College of Dental Sciences and Research, Bhilai, Chhattisgarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402
- [Background] Cortellini P, Pini Prato G, Tonetti MS. Periodontal regeneration of human infrabony defects. II. Re-entry procedures and bone measures. J Periodontol. 1993 Apr;64(4):261-8. doi: 10.1902/jop.1993.64.4.261. PMID 8483088
- [Background] Cortellini P, Pini Prato G, Tonetti MS. Periodontal regeneration of human infrabony defects. I. Clinical measures. J Periodontol. 1993 Apr;64(4):254-60. doi: 10.1902/jop.1993.64.4.254. PMID 8483087
- [Background] Camelo M, Nevins ML, Lynch SE, Schenk RK, Simion M, Nevins M. Periodontal regeneration with an autogenous bone-Bio-Oss composite graft and a Bio-Gide membrane. Int J Periodontics Restorative Dent. 2001 Apr;21(2):109-19. PMID 11829385